CLINICAL TRIAL: NCT06632873
Title: Therapeutic Efficiency and Response to 177Lu-TATE-RGD in Patients With SSTR2 and Integrin αVβ3 Positive Tumors
Brief Title: 177Lu-TATE-RGD in Patients With SSTR2 and Integrin αVβ3 Positive Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Zhu, Clinical Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-TR-II
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: SSTR2 and Integrin αVβ3 Positive Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1.48-3.33 GBq of 177Lu-TATE-RGD (Experimental): The patients were intravenously injected with the dose about 1.48-3.33 GBq(60-100m Ci) 177Lu-TATE-RGD and underwent 68Ga-TATE-RGD PET/CT scans before and after the treatment.
  Interventions: Drug: 177Lu-TATE-RGD

INTERVENTIONS:
Drug: 177Lu-TATE-RGD — accepted intravenous injection of 177Lu-TATE-RGD

SUMMARY:
Researchers has conducted extensive research on the treatment of neuroendocrine tumors with 177Lu-EB-TATE and the treatment of FAP-expressing tumors with 177Lu-EB-FAPI, and some researches have revealed 68Ga-TATE-RGD in imaging studies of neuroendocrine tumors to find that the dual-targeted tracer showed an increasing TBR, suggesting the tracer kinetic advantage of TATE-RGD; compared to the single-target tracer DOTATATE, the dual-target TATE-RGD probe has a clear advantage in detecting liver metastases of NETs, and it can be explored for potential therapeutic uses of TATE-RGD in future studies and used for related companion diagnostics in targeted radioisotope therapy (RLT).

DETAILED DESCRIPTION:
Integrin αvβ3 is highly expressed in certain tumor cells and newly formed blood vessels, making it an ideal target for diagnosis and treatment of integrin αVβ3 positive tumors. 177Lu-TATE-RGD is a novel drug developed independently in China, providing an effective target for the treatment of integrin αVβ3 positive tumors. All patients underwent whole-body 68Ga-TATE-RGD PET/CT screening within one week and received a single intravenous injection of 1.48-3.33 GBq (40-100 mCi) 177Lu-TATE-RGD within one week. Blood samples were collected from the vein in 1-2 mL volumes at 5 minutes, 3 hours, 24 hours, 72 hours, and 168 hours after injection to measure radioactivity. Then, whole-body planar and SPECT/CT imaging was performed at 3, 24, 48, 72, 96, 120, and 168 hours after the injection of 177Lu-TATE-RGD. The in vivo radiation dose of 177Lu-TATE-RGD was analyzed and calculated, and the therapeutic effect and response were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with clear pathological diagnosis and ineffective or progressing clinical conventional treatment;
* tumor lesions with high SSTR2 and RGD untake confirmed on 68Ga-TATE-RGD PET/CT within one week before the injection of 177Lu-TATE-RGD;
* signed written consent.

Exclusion Criteria:

* the exclusion criteria were a serum creatinine level of more than 150 μmol per liter, a hemoglobin level of less than 10.0 g/dl, a white-cell count of less than 4.0× 109/L, a platelet count of less than 100 × 109/L, a total bilirubin level of more than 3 times the upper limit of the normal range and a serum albumin level of more than 3.0 g per deciliter, cardiac insufficiency including carcinoid heart valve disease, a severe allergy or hypersensitivity to radiographic contrast material, claustrophobia;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
StandarStandardized uptake value of 177Lu-TATE-RGD in normal organs and tumors. | through study completion, an average of half-year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value at each time point in normal organs and tumors will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 2 months
  Adverse events within 2 months after the injection and scanning of patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China